CLINICAL TRIAL: NCT05919654
Title: Clinical Evaluation of MyoCare in Europe (CEME): Study Protocol for a Prospective, Multicenter, Randomized, Double-blinded, and Controlled Clinical Trial.
Brief Title: Clinical Evaluation of MyoCare in Europe (CEME)
Acronym: CEME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Cooperativa de Ensino Superior, Politécnico e Universitário (Other); Novovision (Unknown); Instituto de Cirugia Ocular (Other); Miranza Virgen de Lujan (Unknown); ICQO Instituto Quirúrgico de Oftalmología (Unknown); CPO Clinica Privada de Oftalmologia, S.A. (Unknown); Carl Zeiss Vision International GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCM-MIOPIA-01; 2022-001696-14 (EudraCT Number); 22/384-EC_P (Other: CEIm Hospital Clínico San Carlos)
Record Dates: First submitted 2023-05-31; First posted 2023-06-26 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-06

CONDITIONS: Myopia, Progressive
Keywords: myopia
MeSH Terms: conditions — Myopia, Degenerative; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Myocare
  Interventions: Device: MyoCare
- Control (Active Comparator): Clearview
  Interventions: Device: ClearView

INTERVENTIONS:
Device: MyoCare — Children assigned to the study group will wear ZEISS MyoCare lenses, while those assigned to the control group will wear conventional ZEISS ClearView single-vision lenses in their spectacles. Both lenses will be made of the same material (MR8) and hard as well as anti-reflection coating (ZEISS DuraVision Platinum) and will have the same surface treatments.
  Arms: Treatment
Device: ClearView — Children assigned to the study group will wear ZEISS MyoCare lenses, while those assigned to the control group will wear conventional ZEISS ClearView single-vision lenses in their spectacles. Both lenses will be made of the same material (MR8) and hard as well as anti-reflection coating (ZEISS DuraVision Platinum) and will have the same surface treatments.
  Arms: Control

SUMMARY:
A 2-year prospective, multicenter, randomized controlled, and double-blind clinical trial is used to investigate the efficacy of a new design of ophthalmic lenses to slow the progression of myopia. 300 children aged from 6 to 13 years old will be recruited and randomly assigned to a study or control group. The study group will be composed of 150 children wearing MyoCare while the control group will be composed of 150 children wearing Clearview. The inclusion criteria will be myopia with a spherical equivalent between -0.75D and -5.00D, astigmatism < 1.50D, and anisometropia < 1.00D, as well as having a historical evolution of at least -0.50 The primary outcome is to compare the mean annual progression of the spherical equivalent between both groups. The secondary outcomes are axial length, choroidal thickness, phorias, and accommodative status of both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-13 years
* Caucasian ethnicity
* Monocular/binocular decimal visual acuity with correction ≥ 1.00
* Spherical equivalent between -0.75D and -5.00D
* Astigmatism < 1.50D
* Anisometropia < 1.00D
* Evolution of at least -0.50D in one year

Exclusion Criteria:

* Presence of ocular pathology or a history of ocular and systemic abnormalities
* Strabismus or binocular vision problems
* History of eye surgery
* Having previously used some method to control myopia.
* Having contraindications for the application of drugs for cycloplegia/corneal anesthesia

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective refraction | 2 years
  Objective refraction will be taken after cycloplegia as the mean of 3 measurements with the i.profiler (Carl Zeiss Meditec AG, Jena, Germany) autorefractometer. The mean annual progression of the objective refraction will be compared between myopic children treated with ZEISS MyoCare lenses and those who wear a conventional single-vision lens.

SECONDARY OUTCOMES:
Axial length | 2 years
  1. To compare the mean annual progression of axial length between myopic children treated with ZEISS MyoCare lenses and those who wear a conventional single-vision lens.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alvarez-Peregrina C, Sanchez-Tena MA, Martinez-Perez C, Villa-Collar C; Clinical Evaluation of MyoCare in Europe -the CEME Study Group; Ohlendorf A. Clinical Evaluation of MyoCare in Europe (CEME): study protocol for a prospective, multicenter, randomized, double-blinded, and controlled clinical trial. Trials. 2023 Oct 17;24(1):674. doi: 10.1186/s13063-023-07696-0. PMID 37848908